CLINICAL TRIAL: NCT01361516
Title: Comparison of General Anaesthesia and Sedation on the Stone Fragmentation Efficacy of the Third Generation Lithotriptor
Brief Title: Comparison of General Anaesthesia and Sedation on the Stone Fragmentation in Lithotripsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr Saifi Fayez, Hadassah Medical Organisation
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 021711-HMO-CTIL
Record Dates: First submitted 2011-05-11; First posted 2011-05-26 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-04

CONDITIONS: Urolithiasis
Keywords: Urolithiasis; ESWL; Stone Fragmentation efficacy; Sedation; General Anaesthesia
MeSH Terms: conditions — Urolithiasis | interventions — Anesthesia; Lithotripsy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravenous sedation, General anaesthesia (Experimental): IV sedation-ESWL under spontaneous respiration GA - ESWL under controlled respiration
  Interventions: Other: Anaesthesia and Lithotripsy

INTERVENTIONS:
Other: Anaesthesia and Lithotripsy — The efficacy of stone fragmentation during lithotripsy procedure is compared under two types of anaesthesia

SUMMARY:
The aim of the study is to compare the impact intravenous sedation versus general anesthesia on the efficacy of stone fragmentation in extracorporeal shock wave lithotripsy treatment.

DETAILED DESCRIPTION:
The newer lithotriptors were reported to be less efficacious than the Dornier HM3 lithotriptor; and it is not clear the reason why there is decrease in efficacy of the new lithotriptors. Is it due to their small focal point or to increased patient movement while under intravenous sedation.When the patients get sedated then it will be difficult to control their respiratory movements. Retrospective comparisons suggest that intravenous may facilitate earlier discharge if no manipulation of the airway was done; but they are often associated with pain, hypoxemic respiratory episodes and disruptive movements during lithotripsy Instead of intravenous sedation, general anesthesia offer pain free procedures, no movement of the patient and controlled movement of the respiration leads to stable position of the urinary stones and receives persistent shock wave energy on to the stone bringing about better and early fragmentation. Hence we work on the hypothesis that the new generation shock wave lithotripters have a small focal point, every movement of the stone during the respiration or patient movement, will take the stone out of the focus and there results in loss of shocks leading to lithotripsy failure and use of more fluoroscopy for refocusing the stone.

Thus we think the proper choice of anesthetic technique will improve the efficacy of stone fragmentation in shock wave lithotripsy treatment at least in those who are obese and suffers from occult sleep- apnoea syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Renal or upper ureteral stone of less than 2cm
2. A.S.A Grade 1.2.3
3. Age above 18 years

Exclusion Criteria:

1. Mid or lower ureteral stones
2. Bilateral renal stones
3. Multiple stones
4. Use of regional anesthesia
5. Coagulopathies (thrombocytopenia, anticoagulation drugs)
6. Suspected or documented difficult intubation
7. History of chronic opioid abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Measurement of stone fragmentation during lithotripsy treatment under general anesthesia and sedation | One year
  Stone fragmentation is measured as disappearence of the stone on flouroscopic monitoring and number of shocks utilised to break the stone during the lithotripsy treatment under general anesthesia (controlled ventilation) or with intravenous sedation(spontaneous ventilation)will be compared in this study.

SECONDARY OUTCOMES:
Anesthesia complications | One year
  We are going to measure pain score (VAS 0-10)and postoperative hypoxemia, saturation below 90% well be considered as hypoxemic event

CONTACTS AND LOCATIONS:
Overall Officials: Fayez Saifi, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel